CLINICAL TRIAL: NCT01980836
Title: The Effect of Tocilizumab on the Cellular Immune Response to Seasonal Influnza Vaccine in Patients With Rheumatoid Arthritis
Brief Title: Effect of Tocilizumab to the Cellular Immune Response to Influenza Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-13-OE-245-CTIL
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Rheumatoid Arthritis; Cellular Immune Response
Keywords: Rheumatoid arthritis; Tocilizumab; Seasonal influenza vaccine
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seasonal influenza vaccine in tocilizumab treated RA patients (Active Comparator): RA patients treated with tocilizumab
  Interventions: Biological: Seasonal influenza vaccine
- Seasonal influenza vaccine to Healthy controls (Active Comparator): Healthy controls will be vaccinated against seasonal influenza
  Interventions: Biological: Seasonal influenza vaccine

INTERVENTIONS:
Biological: Seasonal influenza vaccine

SUMMARY:
Patients with rheumatoid arthritis (RA) are prone to respiratory infections and therefore recommmended to receive vaccination against seasonal influenza. We and others have shown a relatively preserved humoral response to vaccination in RA patients. However, the cellular response as well as the effect of biologics such as tocilizumab on the cellular response has not been weel studied. The purpose of this study is the evaluate the effect of tocilizumab on the cellular immune response to influenza vaccine in patients with RA in comparison with healthy controls

DETAILED DESCRIPTION:
Inclusion criteria :

* RA patients
* Above the age of 18
* Treated with tocilizumab at least 3 months

Exclusion criteria:

-egg allergy

Design of the study :

- Patients and controls will be vaccinated against sesaonal influenza. Blood will be taken the day of vaccination and 4 weeks after.

PBMC isolation The PBMCs will bere isolated from heparinized venous blood by density gradient centrifugation on Lymphoprep (Axis-Shield, Oslo, Norway) immediately after blood was drawn. The cells will be counted and suspended in RPMI 1640 supplemented with heat-inactivated 10% fetal calf serum, penicillin 100U/ml, streptomycin 0.1 mg/ml, and 2 mM L-glutamine (Biological Industries, Israel).

IFN-gamma secretion from PBMCs IFN-gamma secretion levels will be measured by ELISA in the supernatants of PBMCs that will be stimulated with either an influenza antigen mixture or with SEB, or left untreated.

Granzyme B activity assay The PBMCs will be cultured at 0.5 ml/well in 48-well plates (1.8X106 cells/well) and stimulated with an influenza antigen mix and SEB as described above. The cells will be lysed in lysis buffer (150mM NaCl, 15mM Tris, 1% Triton x100), then stored at

-760C. Granzyme B activity will be measured according to the protocol described by Gijzen et al. [13]. Briefly, frozen cell lysates will be subjected to three freeze/thaw cycles to enable the release of Granzyme B. Recombinant Granzyme B standards (Enzo Life Sciences International, Inc., PA) and cell lysates will be added in duplicate to a 96-well plate (20 µl/well). The reaction will start upon the addition of 80 μl of substrate solution containing 400 μM of Ac-IEPD-pNA substrate (Calbiochem, Darmstadt, Germany) in assay buffer (100mM HEPES pH 7.5, 10% (w/v), sucrose, 0.1% (w/v) CHAPS, and 10 mM DTT (Sigma Aldrich, Rehovot, Israel). The plate will be sealed, covered and incubated in a dark humidified chamber at 370C for 20 h. After incubation, the plate will be read at 405 nm. Granzyme B units will be calculated using a 4th order polynominal curve with a log (concentration)-log (absorbance) plot, and corrected for protein concentrations by the BCA protein assay (Thermo Scientific, IL).

The humoral response The antibody response will be measured by the HI test according to a standard WHO procedure as previously described [14]. The titer of an antiserum not showing any inhibition will be recorded as 1/10. Humoral response is defined as either a fourfold or greater rise in the titer of HI antibodies, or a rise from a non-protective baseline level (<1/40) to 1/40). Geometric mean titers of antibodies wull be calculated to assess the immunity of the whole group.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis patients treated with Tocilizumab for at least 3 months
* Above the age of 18

Exclusion Criteria:

* Allergy to eggs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Cellular response | 4 weeks
  As described in the study design using the Interferin gamma and granzyme B levels

SECONDARY OUTCOMES:
Humoral response | 4 weeks
  Using an hemaglutination inhibition test as described in the study design

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Elkayam O, Amir S, Mendelson E, Schwaber M, Grotto I, Wollman J, Arad U, Brill A, Paran D, Levartovsky D, Wigler I, Caspi D, Mandelboim M. Efficacy and safety of vaccination against pandemic 2009 influenza A (H1N1) virus among patients with rheumatic diseases. Arthritis Care Res (Hoboken). 2011 Jul;63(7):1062-7. doi: 10.1002/acr.20465. PMID 21425247
- [Background] Arad U, Tzadok S, Amir S, Mandelboim M, Mendelson E, Wigler I, Sarbagil-Maman H, Paran D, Caspi D, Elkayam O. The cellular immune response to influenza vaccination is preserved in rheumatoid arthritis patients treated with rituximab. Vaccine. 2011 Feb 11;29(8):1643-8. doi: 10.1016/j.vaccine.2010.12.072. Epub 2011 Jan 4. PMID 21211590